CLINICAL TRIAL: NCT03615092
Title: Acellular Dermal Matrix Graft In Root Coverage of Gingival Recessions With Previously Restored Cervical Lesions. A Controlled Clinical Trial
Brief Title: Acellular Dermal Matrix Graft In Root Coverage of Gingival Recessions With Previously Restored Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Phd, Ms, DDs. Chairman of Periodontolgy, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 0002.0.138.000.-11
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Gingival Recession
Keywords: Acellular dermal matrix graft; Clinical Trial; Root coverage; Noncarious cervical lesion
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Controlled Split-mouth clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinical parameters were screened by one single examiner that was not aware of the procedures
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- Test Group (Active Comparator): Active Comparator: gingival recession with a previous restored cervical lesion
  the aim of this study is to compare if the acellular dermal matrix graft is as efficient as a substitute for the connective graft used in root coverage of gingival recessions with non carious cervical lesions.
  Interventions: Procedure: Root coverage with extended flap technique and acelular dermal matrix
- Control Group (Placebo Comparator): the aim of this study is to compare if the acellular dermal matrix graft is as efficient as a substitute for the connective graft used in root coverage of gingival recessions with non carious cervical lesions. The control group had no cervical lesion, and was treated with the same technique as the acelular dermal matrix graft
  Interventions: Procedure: Root coverage with extended flap technique and acelular dermal matrix

INTERVENTIONS:
Procedure: Root coverage with extended flap technique and acelular dermal matrix — At one side, the root coverage have been done with a extended flap technique and acellular dermal matrix and there was no cervical lesion. At the other side, the same technique was performed, but the gingival recession was associated with a noncarious cervical lesion.

SUMMARY:
Patients with high standards of oral hygiene frequently search for buccal gingival recession (GR) treatment due to cervical wear, root sensitivity and compromising aesthetics. The cervical lesion (NCCL) is commonly produced by improper toothbrushing techniques, sharing the same etiology of GR. Many different surgical approaches have been described. The association of a graft to the coronally advanced flap had demonstrated the best long-term outcome for root coverage. But, substitutes for the autogenous graft must be studied. Therefore, the aim of this clinical trial was to investigate the effectiveness of the acellular dermal matrix graft (ADMG) in root coverage associated with a previous restored cervical lesion or not.

Material and methods: Seventeen individuals with bilateral GR were included in the study. At one side, the GR must present a previously restored cervical lesion, as the test group (TG). The contralateral arch, must present GR with an intact root surface (CG). All patients were treated with the extended flap technique associated with the ADMG. All clinical parameters were assessed at baseline and 6-months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* CEJ without significant damage;
* localized bilateral RT112 gingival recession ≥3 mm in the same arch, in which one had a non-carious cervical lesion (NCCL) restored with composite and the opposite one was intact

Exclusion Criteria:

* previous periodontal surgical treatment on the involved sites;
* smokers
* pregnants or lactating
* compromised systemic health and contraindications for periodontal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-01-30 (Actual); Primary Completion 2011-10-05 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Root coverage | 6 months
  Root coverage is measured by the difference between the gingival recession height at 6 months and baseline

SECONDARY OUTCOMES:
Keratinized tissue | 6months
  The difference between keratinized tissue width and depth at 6 months and at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry of Ribeirao Preto - University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No